CLINICAL TRIAL: NCT01440465
Title: Management of Nausea and Vomiting Chemotherapy-induced in Normandy
Acronym: NAVI
Status: Completed | Type: Observational
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Other Study IDs: NAVI
Record Dates: First submitted 2011-09-15; First posted 2011-09-26 (Estimated); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Cancer; Nausea; Vomiting
Keywords: chemotherapy; cancer; nausea; vomiting
MeSH Terms: conditions — Neoplasms; Nausea; Vomiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objective of this study was to evaluate the various parameters involved in the occurrence of nausea / vomiting during the first cycle of chemotherapy for solid tumors or hematologic among a group of chemotherapy-naive patients, despite anti standardized-emetics protocols.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years
* With solid tumors or hematologic in first line chemotherapy, administered intravenously,
* Able to understand the meaning of the questions
* Having given their written consent to participate in the survey.

Exclusion Criteria:

This does not concern patients who:

* Do not give their consent for participation
* Do not speak French
* Suffer from cognitive deficits
* Are under therapy
* Must receive a combination of radio-chemotherapy
* Present an occlusive syndrome
* Metastases (s) brain (s) clinically symptomatic (s) or radiologically proven (s) or a (of) tumor (s) brain (s)
* Have been previously treated with chemotherapy
* Present a cons-indication to corticosteroids, with anti-serotonin or NK1 receptor inhibitors
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with first line chemotherapy with intravenous (IV) to solid tumors or hematologic.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-07; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JOLY Florence, Pr, Principal Investigator — Centre François Baclesse
Locations (6):
- France (6):
  - Centre de la Baie, Avranches
  - Centre hospitalier, Bayeux
  - Centre Maurice Tubiana, Caen
  - Centre François Baclesse, Caen
  - Centre hospitalier public du cotentin, Cherbourg-Octeville
  - Centre Jacques Monod, Flers

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible patients were older than 18 years, chemotherapy naive, and with a histologically proven solid malignant tumour requiring chemotherapy whatever the stage of the disease.
  Patients had to understand the procedures and agree to participate in the study by giving written informed consent.
Groups:
- Experimental arm: Chemotherapy-naïve patients are included during the first cycle of treatment to assess frequency and intensity of chemotherapy-induced nausea and vomiting.
Period: Overall Study
Arm/Group | Experimental arm
Started | 300
Completed | 291
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Experimental Arm
Number analyzed (Participants) | 291
Age, Continuous [Median (Full Range); unit: years] | 57 [24 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 248
  Male | 43
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Stage of the disease [Count of Participants; unit: Participants] — Participants were categorized according to the clinical treatment setting at the time of inclusion, which reflects disease severity and treatment intent. Three clinical categories were defined:
  Adjuvant setting: patients with resected disease receiving postoperative systemic therapy with curative intent.
  Neoadjuvant setting: patients receiving systemic therapy prior to planned tumor resection with curative intent.
  Metastatic setting: patients with unresectable or metastatic disease receiving systemic therapy with palliative intent.
  Participants
    Adjuvant setting | 219
    Neo-adjuvant setting | 27
    Metastatic setting | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Nausea and Vomiting
Description: acute nausea and vomiting and/or delayed measured by the tool of anti emetic MAT MASCC. Such self-administered questionnaire was found to be sensitive to detect the different dimensions of chemo-induced nausea and vomiting and to perform well against a daily assessment of nausea and vomiting. The MAT questionnaire separately asks for acute (within 24h of initial administration of chemotherapy) and delayed (from 24h to 4 days after chemotherapy) chemo-induced nausea and vomiting by asking the patient to fill out the first page the day after chemotherapy referring to the first 24h following chemotherapy and the second page 4 days after chemotherapy concerning the period from the day after to 4 days after chemotherapy. Clinically significant nausea was defined by reported nausea intensity >=3 on a 0-10 scale, 10 being the highest intensity of nausea. Clinically significant chemo induced nausea/vomiting was defined by greater than or equal to one nausea episode/vomiting, respectively.
Time Frame: 24 hours
Population: Data from MAT to measure chemotherapy-induced nausea and vomiting were available for 248 patients of the 291 included (85.2%).
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental arm
Number analyzed (Participants) | 248
Participants | 101

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 6 months
Arm/Group | Experimental arm
All-Cause Mortality (participants affected / at risk) | 1/291
Serious Adverse Events (participants affected / at risk) | 1/291
Other Adverse Events (participants affected / at risk) | 260/291
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental arm (N=291)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental arm (N=291)
NAUSEA (GASTROINTESTINAL DISORDERS) | 156 (211)
ABDOMINAL PAIN (GASTROINTESTINAL DISORDERS) | 3 (4)
ASCITES (GASTROINTESTINAL DISORDERS) | 1 (1)
PLEURAL EFFUSION (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 (1)
HEPATIC CYTOLYSIS (HEPATOBILIARY DISORDERS) | 1 (1)
MUCOSAL INFLAMMATION (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 16 (16)
FEBRILE NEUTROPENIA (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 12 (12)
MALAISE (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 3 (3)
ABDOMINAL PAIN UPPER (GASTROINTESTINAL DISORDERS) | 7 (7)
MYALGIA (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 4 (4)
VOMITING (GASTROINTESTINAL DISORDERS) | 28 (34)
BRONCHITIS (INFECTIONS AND INFESTATIONS) | 3 (3)
HEADACHE (NERVOUS SYSTEM DISORDERS) | 16 (17)
INSOMNIA (PSYCHIATRIC DISORDERS) | 3 (3)
APLASIA (CONGENITAL, FAMILIAL AND GENETIC DISORDERS) | 2 (2)
PYELONEPHRITIS (INFECTIONS AND INFESTATIONS) | 1 (1)
ANGINA PECTORIS (CARDIAC DISORDERS) | 2 (2)
ESCHERICHIA INFECTION (INFECTIONS AND INFESTATIONS) | 1 (1)
PYREXIA (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 13 (13)
RASH (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1 (1)
FUNGAL INFECTION (INFECTIONS AND INFESTATIONS) | 2 (2)
FOLLICULITIS (INFECTIONS AND INFESTATIONS) | 2 (2)
ALOPECIA (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 44 (44)
NEUROPATHY PERIPHERAL (NERVOUS SYSTEM DISORDERS) | 14 (14)
ASTHENIA (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 36 (36)
DECREASED APPETITE (METABOLISM AND NUTRITION DISORDERS) | 4 (4)
VAGINAL INFECTION (INFECTIONS AND INFESTATIONS) | 1 (1)
FEBRILE BONE MARROW APLASIA (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 3 (3)
VISUAL IMPAIRMENT (EYE DISORDERS) | 1 (1)
MIGRAINE (NERVOUS SYSTEM DISORDERS) | 7 (7)
HERPES ZOSTER (INFECTIONS AND INFESTATIONS) | 1 (1)
BONE PAIN (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 4 (4)
TREMOR (NERVOUS SYSTEM DISORDERS) | 2 (2)
THROMBOCYTOPENIA (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 2 (2)
NEUTROPENIA (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 16 (19)
SCIATICA (NERVOUS SYSTEM DISORDERS) | 1 (1)
TOOTH ABSCESS (INFECTIONS AND INFESTATIONS) | 1 (1)
CONSTIPATION (GASTROINTESTINAL DISORDERS) | 3 (3)
DRY SKIN (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 2 (2)
SINUSITIS (INFECTIONS AND INFESTATIONS) | 2 (2)
ACUTE KIDNEY INJURY (RENAL AND URINARY DISORDERS) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 (1)
ANAEMIA (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 9 (9)
PARAESTHESIA (NERVOUS SYSTEM DISORDERS) | 4 (4)
DIARRHOEA (GASTROINTESTINAL DISORDERS) | 13 (13)
NASOPHARYNGITIS (INFECTIONS AND INFESTATIONS) | 4 (4)
NECK PAIN (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 (1)
HYPERSENSITIVITY (IMMUNE SYSTEM DISORDERS) | 1 (1)
APHTHOUS ULCER (GASTROINTESTINAL DISORDERS) | 3 (3)
PALPITATIONS (CARDIAC DISORDERS) | 1 (1)
PHARYNGITIS (INFECTIONS AND INFESTATIONS) | 2 (2)
ARTHRALGIA (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (GASTROINTESTINAL DISORDERS) | 2 (2)
TOOTHACHE (GASTROINTESTINAL DISORDERS) | 2 (2)
ANXIETY (PSYCHIATRIC DISORDERS) | 2 (2)
INTESTINAL ISCHAEMIA (GASTROINTESTINAL DISORDERS) | 1 (1)
PAIN (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 4 (4)
BACK PAIN (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 3 (3)
ORAL CANDIDIASIS (INFECTIONS AND INFESTATIONS) | 1 (1)
PRURITUS (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1 (1)
DENTAL CARE (SURGICAL AND MEDICAL PROCEDURES) | 1 (1)
HOT FLUSH (VASCULAR DISORDERS) | 1 (1)
DYSPHAGIA (GASTROINTESTINAL DISORDERS) | 2 (2)
BLOOD GLUCOSE INCREASED (INVESTIGATIONS) | 1 (1)
HYPERTHERMIA (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 1 (1)
HYPOTENSION (VASCULAR DISORDERS) | 2 (2)
URINARY TRACT INFECTION (INFECTIONS AND INFESTATIONS) | 2 (2)
DYSAESTHESIA (NERVOUS SYSTEM DISORDERS) | 1 (1)
COUGH (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 2 (2)
GASTROENTERITIS (INFECTIONS AND INFESTATIONS) | 2 (2)
HAEMORRHOIDS (GASTROINTESTINAL DISORDERS) | 1 (1)
EPISTAXIS (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 (1)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1 (1)
CANDIDIASIS (INFECTIONS AND INFESTATIONS) | 1 (1)
GENERAL PHYSICAL HEALTH DETERIORATION (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 1 (1)
LARYNGITIS (INFECTIONS AND INFESTATIONS) | 1 (1)
FATIGUE (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 3 (3)
TOOTH INFECTION (INFECTIONS AND INFESTATIONS) | 1 (1)
TACHYCARDIA (CARDIAC DISORDERS) | 1 (1)
OROPHARYNGEAL CANDIDIASIS (INFECTIONS AND INFESTATIONS) | 1 (1)
VULVOVAGINAL MYCOTIC INFECTION (INFECTIONS AND INFESTATIONS) | 1 (1)
MUSCLE SPASMS (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 (1)
ODYNOPHAGIA (GASTROINTESTINAL DISORDERS) | 1 (1)
WEIGHT DECREASED (INVESTIGATIONS) | 1 (1)
DYSGEUSIA (NERVOUS SYSTEM DISORDERS) | 1 (1)
CHILLS (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No